CLINICAL TRIAL: NCT03281031
Title: Diagnostic Performance of MRI as an Alternative to CT Following a Non-diagnostic Ultrasonography in Young Women With Acute/Subacute Abdominal Pain : a Prospective Multicenter Study
Brief Title: MRI as an Alternative to CT for Exploration of Acute Abdominal Pain in Young Women
Acronym: IRMADA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UF9803; 2017-A00725-48 (Other: Agence Nationale de Sécurité des Médicaments France)
Record Dates: First submitted 2017-07-27; First posted 2017-09-13 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2021-12

CONDITIONS: Acute Abdominal Pain; Pelvic Pain
Keywords: MRI; Acute abdominal pain; Pelvic pain; Diagnostic performance; Young women
MeSH Terms: conditions — Abdomen, Acute; Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional MRI Examination (Other): Single arm, all patient will undergo CT followed by additional MRI examination
  Interventions: Procedure: Additional MRI Examination

INTERVENTIONS:
Procedure: Additional MRI Examination — MRI will be performed using a short protocol within 6 hours from CT and with blinding from CT results

SUMMARY:
Objective :

To demonstrate diagnostic performances of Magnetic Resonance Imaging (MRI) as compared to Computed Tomography (CT) as a second intention imaging modality in young women with acute non traumatic abdominopelvic pain and non contributive ultrasonography.

DETAILED DESCRIPTION:
Methods :

Consecutive women aged 18-40 years old with acute abdominopelvic pain referred to CT by the emergency Physician or gynaecologist after a non contributive ultrasonography will be included.

After obtaining informed consent, all patients will undergo standard CT followed by an additional MRI examination, performed using a short MRI protocol and within 6 hour from CT.

The gold standard or reference diagnosis will be established in consensus by an expert panel at 3 months follow up using a standardized diagnosis form.

A retrospective reading will be performed independently for CT and MRI by radiologists blinded to the reference diagnosis, using the same standardized diagnosis form.

CT and MRI accuracies will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years old
* Women referred to CT following a non contributive ultrasonography
* Women with acute non traumatic abdominopelvic pain (less than 5 day-duration)
* Women with informed consent
* Women with affiliation to health insurance

Exclusion Criteria:

* Women who underwent abdominopelvic surgery in the previous month
* Suspicion of vital emergency such as shock preventing any delayed management caused by MRI examination
* Contra-indication to MRI, including pace maker, ferro-magnetic material, foreign bodies with risk of mobilization during MRI examination
* Women yet included in the study or included in another study
* Women pregnant (positive beta chorionic gonadotrophic hormone testing) or breastfeeding
* Women unable to undergo informed consent (vulnerable or protected by law)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 347 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performances comparison between CT and MRI | 3 months
  Diagnostic performances (sensitivity, specificity, predictive values) comparison between CT and MRI

SECONDARY OUTCOMES:
Diagnostic performances of a conditional imaging strategy including first MRI for all cases and CT in cases where MRI is non contributive | 3 months
  Diagnostic performances (sensitivity, specificity and predictive values) of a conditional imaging strategy including first MRI for all cases and CT in cases where MRI is non contributive (strategy built retrospectively)
Diagnostic performances of unenhanced MRI sequences versus complete MRI examination | 3 months
  Diagnostic performances (sensitivity, specificity and predictive values) of unenhanced MRI sequences versus complete MRI examination (including both unenhanced and enhanced sequences)
Inter-reader agreement for MRI and CT diagnoses | 3 months
  Inter-reader agreement (Kappa statistics) for MRI and CT diagnoses (retrospective reading)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid MILLET, MD, PhD, Principal Investigator — Departement of Medical Imaging - Montpellier University Hospital LAPEYRONIE Hospital
Locations (1):
- Departement of Medical Imaging, Montpellier, France